CLINICAL TRIAL: NCT00942916
Title: Serum Inflammatory Marker in Patients With Diagnosis of Nontuberculous Mycobacterial Pulmonary Infection
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200903008R
Record Dates: First submitted 2009-07-19; First posted 2009-07-21 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-06

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Infection
Keywords: Make sure the difference of the serum inflammatory marker between the two groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with confirmed diagnosis of NTM pulmonary disease: Those with sputum mycobacterial culture yielded the same NTM species for at least two sets within one year.
- Patients with not definite NTM pulmonary disease: Those who had sputum culture yielded NTM but did not satisfy the criteria for diagnosis with NTM pulmonary disease.

SUMMARY:
This study is for those who had nontuberculous mycobacterial pulmonary infection with higher a serum inflammatory marker than those who had colonization.

DETAILED DESCRIPTION:
Nontuberculous mycobacteria (NTM), not like Mycobacterium tuberculosis, is ubiquitous in environment including soil and water. Therefore, NTM pulmonary infection is not diagnosed only by microbiology of respiratory specimen but also clinical and radiographical findings.(1) Due to airway NTM colonization is not uncommon in sputum, diagnosis of pulmonary NTM infection is a big challenge in clinical practice. Especially NTM burden is increasing in recent literature.(2,3) Besides, the short-term mortality is reported higher in patients with NTM infection in medical ICU by Shu et al.(4) Early diagnosis and then treatment of NTM infection become important though NTM infection is considered as indolent process before.(1) Inflammatory marker in the patients with NTM being isolated from respiratory specimens is an indicator for differentiating true infection from colonization.(5,6) Those inflammatory factors might include blood white count, C-reactive protein, cytokines, procalcitonin , trigger receptor expressed on myeloid cell-1 (TREM-1) and Toll-like receptor-2. We therefore conduct this prospective study for analyzing

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years
* study group : Satisfied the criteria for NTM pulmonary disease according to the ATS diagnosis guidelines.
* control groups: they had positive sputum culture for NTM but not fulfilled the diagnosis criteria

Exclusion Criteria:

* Those with bleeding tendency
* No inform consent
* Female with pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was diagnosed as NTM pulmonary disease. They had satisfied at least microbiological, radiographical and clinical criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of NTM pulmonary disease according to the ATS guidelines | 2 year

SECONDARY OUTCOMES:
mortality | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Yun-Lin County, Taiwan